CLINICAL TRIAL: NCT06799026
Title: A Phase 1 Study of Vaccination With Dendritic Cell (DC)/Multiple Myeloma (MM) Fusions in Combination With Elranatamab in Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Avigan (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, David Avigan, Sponsor Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-439
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: MM; Multiple Myeloma; Relapse Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elranatamab + DC/MM Vaccine + GM-CSF (Experimental): * Baseline visit and assessments
  * Leukapheresis
  * Cycle 1 (28-day cycle):
    --Days 1, 8, 15, and 22: Predetermined dose of Elranatamab 1x daily
  * Cycle 2 (28-day cycle):
    --Days 1, 8, 15, and 22: Predetermined dose of Elranatamab 1x daily
  * Cycles 3 through 5 (28-day cycles):
    * Bone marrow biopsy/aspiration prior to first DC/MM fusion vaccine
    * Days 1, 8, 15, and 22: Predetermined dose of Elranatamab 1x daily
    * Day 8: Predetermined doses of DC/MM fusion vaccine 1x daily and GM-CSF 1x daily (GM-CSF for days 9 through 11 are self-administered)
  * Cycle 6 (28-day cycle):
    * Bone marrow biopsy/aspiration on Cycles 6, 9, and 12
    * Days 1, 8, 15, and 22: Predetermined dose of Elranatamab 1x daily
  * Cycle 7 through 12 (28-day cycles):
    * Cycle 7 Day 1 only: Bone marrow biopsy/aspiration
    * Days 1 and 15: Predetermined dose of Elranatamab 1x daily
  * After end of treatment, bone marrow biopsy/aspiration at months 1, 3, and 6
  * 6 month follow up visit
  * Long term follow up 5 years
  Interventions: Drug: Elranatamab; Biological: GM-CSF; Biological: DC/MM Fusion Vaccine

INTERVENTIONS:
Drug: Elranatamab — Bispecific T-cell engager antibody, 1.9 and 1.1 mL vials, via subcutaneous (under the skin) injection per protocol.
  Other Names: PF-06863135; Elranatamab-bcmm; Elrexfio
Biological: GM-CSF — Granulocyte-Macrophage Colony-Stimulating Factor, via subcutaneous (under the skin) injection per protocol.
  Other Names: Granulocyte-Macrophage Colony-Stimulating Factor
Biological: DC/MM Fusion Vaccine — Dendritic Cell and tumor fusion vaccine, via subcutaneous (under the skin) injection per protocol.
  Other Names: Dendritic Cell/Tumor Fusion Vaccine

SUMMARY:
This research is being done to determine if the combination of the Dendritic Cell (DC)/ Multiple Myeloma (MM) fusion vaccine with elranatamab is safe and effective in treating Relapsed or Refractory Multiple Myeloma (MM).

The names of the study drugs and vaccine involved in this study are:

* DC/MM fusion vaccine (a personalized cancer vaccine in which harvested participant tumor cells are fused with harvested participant dendritic blood cells)
* Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) (a type of growth factor)
* Elranatamab (a type of T-cell engager antibody)

DETAILED DESCRIPTION:
This is a phase 1 study to evaluate the feasibility, safety, clinical and immune effects of DC/MM fusion vaccine in combination with Elranatamab in participants with relapsed/refractory multiple myeloma. The DC/MM fusion vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells. This vaccine is individualized for each participant using dendritic cells (type of immune cells) from each participant. GM-CSF contains a substance that helps make more white blood cells. This medication is being used to possibly increase the effectiveness of the DC/MM fusion vaccine.

The U.S. Food and Drug Administration (FDA) has not approved DC/MM fusion vaccine as a treatment for Relapsed or Refractory Multiple Myeloma.

The FDA has not approved GM-CSF as a treatment for Relapsed or Refractory Multiple Myeloma.

The FDA has approved elranatamab as a treatment option for Relapsed or Refractory Multiple Myeloma.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, urine tests, study drug subcutaneous (under the skin) injections, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, and bone marrow biopsies and aspirations (or collections).

Participants will receive study treatment for up to 12 cycles (28-day cycles) and will be followed for up to 5 years.

It is expected that about 25 people will take part in this research study.

Pfizer is funding this research study by providing one of the study drugs, Elranatamab.

ELIGIBILITY:
Inclusion Criteria for Tumor Collection:

* Participants must have an established diagnosis of multiple myeloma
* Participant must have multiple myeloma and have relapsed following or are refractory to proteasome inhibitors, IMiDs and anti-CD38 mAb therapy
* Participants must have at least 3 prior lines of therapy
* Participants must be ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Participants must have > 20% plasma cells in the bone marrow core or aspirate differential <30 days prior to enrollment.
* ANC > 1K/uL; Platelets > 50 K/uL without transfusional support
* Participants must have adequate organ function as defined below:

  * Total bilirubin ≤1.5 x institutional upper limit of normal
  * AST ≤ 3 x institutional upper limit of normal
  * ALT ≤ 3 x institutional upper limit of normal
  * Creatinine clearance ≥ 40 mL/min for participants with creatinine levels above institutional normal
* The effects of DC/MM fusion vaccine on the developing human fetus are unknown. For this reason, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier methods of birth control or abstinence) prior to study enrollment and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of treatment.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria for Tumor Collection:

* Patients who are receiving any other investigational agents.
* Patients with purely non-secretory MM [absence of a monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence- Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques and the absence of involved serum free light chain >100 mg/L]. Patients with light chain MM detected in the serum by free light chain assay are eligible.
* Patients with Plasma Cell Leukemia
* Because of compromised cellular immunity, patients who have a known human immunodeficiency virus (HIV), active hepatitis C virus (HCV) or active hepatitis B virus (HBV).
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure (see Appendix H), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening will be documented by the investigator as not medically relevant.
* Active and clinically significant autoimmune or inflammatory disorder requiring active treatment
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Note: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: non- invasive cancer (such as, any in situ cancers) and basal cell or squamous cell carcinoma of the skin.
* Female patients who are pregnant (positive β-HCG) or breastfeeding
* Prior organ transplant requiring immunosuppressive therapy.
* Patients who previously received PD-1 antibody and have experienced toxicities resulting in treatment discontinuation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of GBS or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.

Eligibility Criteria Prior to Vaccination with DC/MM fusions

* Resolution of all elranatamab related ≥ grade 3 or higher toxicities to grade 1 or baseline. Isolated laboratory abnormalities that are not considered to be clinically significant are not exclusionary.
* Successful production of at least 2 vaccines with a minimum of 1 x 106 fusion cells per vaccine
* Absence of disease progression following 2 cycles of elranatamab therapy
* ECOG performance status ≤ 2

Participants must have adequate organ function as defined below:

* Total bilirubin ≤ 1.5 x institutional upper limit of normal
* AST ≤ 3 x institutional upper limit of normal
* ALT ≤ 3 x institutional upper limit of normal
* ANC > 1K/uL; Platelets > 50 K/uL without transfusional support
* Creatinine clearance ≥ 40 mL/min for participants with creatinine levels above institutional normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Administration of DC/MM Vaccine | 1 Year
  Feasibility is defined as number of patients who successfully get vaccine
Grade 3-4 Non-hematologic Rate | 1 Year
  Grade 3-4 non-hematologic Rate is defined as the percentage of participants who experienced a maximum grade 3/4 non-hematologic based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Grade 3-4 hematologic Rate | 1 Year
  Grade 3-4 hematologic Rate is defined as the percentage of participants who experienced a maximum grade 3/4 hematologic based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | 18 months
  Overall survival based on the Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Median Progression Free Survival (PFS) | 1 Year
  PFS based on Kaplan Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation.
Elranatamab Toxicity Rate | 1 Year
  Elranatamab Toxicity Rate is defined as percentage of participants who experienced elranatamab toxicity including cytokine release syndrome, neurotoxicity and infections based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
MRD Negative Disease Rate at 1 Year | 1 Year
  MRD Negative Disease Rate at 1 Year is defined as the percentage of participants who are MR- negative after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu